CLINICAL TRIAL: NCT01992419
Title: Evaluation of Cardiac Arrest Recognition by Non-physicians Dispatchers in the Paris Fire Brigade Emergency Call Dispatch Center
Brief Title: Evaluation of Out-of-Hospital Cardiac Arrest Recognition by Non-physicians Dispatchers in a French Emergency Dispatch Call Center
Acronym: OCAR
Status: Completed | Type: Observational
Sponsor: Fire Brigade Of Paris Emergency Medicine Dept (Other)
Responsible Party: Principal Investigator, Dr Jost D., Medical Doctor, responsible for clinical research at Paris Fire Brigade, Fire Brigade Of Paris Emergency Medicine Dept
Other Study IDs: bspp2013
Record Dates: First submitted 2013-11-07; First posted 2013-11-25 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Out-of-hospital Cardiac Arrest
Keywords: Out-of-hospital Cardiac arrest; telephone dispatch assisted resuscitation; cardiac arrest phone detection
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to measure an improvement in the detection rate of cardiac arrest (CA) in the Dispatch Center as a result of debriefings and repeated trainings for non-medical operators who receive emergency calls.

DETAILED DESCRIPTION:
1. . Justification

   The performance of phone-guided chest compressions is recommended to minimize the No Flow risk (1). Pre-arrival instructions and dispatch-assisted chest compressions are the first link in the chain of survival, determining the effectiveness of subsequent links. This first link is only possible if a prior detection of cardiac arrest was made.

   The Dispatch Center of the Fire Brigade of Paris receives more than 7,000 calls per day, including 8-10 calls for cardiac arrest. The establishment of specific training and experience feedback with emergency dispatchers should improve the detection of cardiac arrest (CA) by the same dispatchers.
2. . Objectives

   The main objective is to measure an improvement in the detection rate of CA in the Dispatch Center as a result of debriefings and repeated trainings for non-medical operators who receive emergency calls.

   The secondary objective is to identify risk factors for CA non-detection by those emergency dispatchers.
3. . Materials and Methods

   Experimental design:

   Observational prospective non-randomized controlled study. Type "before and after" study. Three observation periods are defined over a total period of 20 months.

   Different actions before and during each period:

   Period 1 Period 2 Period 3 Algorithm available to emergency dispatchers + + + New algorithm - - + Basic training for new operators - + + Daily briefing +/- +/- + Systematic Debreafing - - + Specific course before period - - + Table leaders training - - + Heads of room training - - +

   Period 1 is preceded and accompanied by the diffusion of a decision algorithm available to emergency dispatchers

   Period 2 is accompanied by:
   * Short briefings, twice daily, in the presence of operators on duty that day
   * Debriefing immediately after the call with some operators (but not systematically, depending on their availability).

   Period 3 is preceded by information to the Dispatch Center managers (heads of room and table leaders) and a short course about detection of CA (1 hour) for all operators. During this same period, a daily briefing for operators is established.

   The study is based on the three CA call periods' audio recordings

   For each period, all calls related to CA on the field were listened to and evaluated.

   Each call had a double audition:
   * one audition by an instructor, responsible for managing calls in the Dispatch Center, and
   * one audition by two emergency physicians experienced in the management of emergency calls.

   The second listening physician helped to verify, correct, and complete the variables collected during the first listening

   The variables collected during listening were:
   * "detectability of the CA"
   * detection or not of the CA
   * the causes of non-detection
   * the occurrence of dispatch-assisted chest compression
   * the time between the start of the call and the time the operator pronounces the words "cardiopulmonary Resuscitation" or "CPR" or "chest compressions"
   * the time between the start of the call and the first real chest compression
   * causes for non-realization of chest compressions
   * the presence or absence of a public defibrillator

   Other variables collected - Variables corresponding to the Utstein style:
   * Epidemiological variables (age, sex, location, background)
   * Specific backup system variables: time alert - use of an AED
   * Specific first aid and medical management variables:

     * type of rhythm detected by AED on the arrival of rescuers
     * Success of first AED's shock (loss of ventricular fibrillaton (VF)5 seconds after shock)
     * Number of shocks administered by the AED in the first 10 minutes of support by rescuers
     * Recovery of a palpable pulse in the presence of rescuers, before the arrival of the medical team
     * Resuscitation undertaken by the medical team YES/NO
     * Injection of adrenaline: YES/NO
     * Transport to the hospital with beating heart: YES/NO
     * Released resuscitation YES/NO
     * Survival to one year after the CA
     * Quality of survival (CPC score) at 6 months, 1 year

   Main judgment criteria:
   * Detection of CA by the emergency dispatcher:

     * Detection is considered positive if the dispatcher formalized the presence of a CA , either on the software, or orally with the words "CPR" or "chest compression" at any time during the recorded call.
     * It is considered negative if the dispatcher never suggested, neither orally nor in writing, the possibility of the presence of a CA.
   * Secondary endpoints:

     * Median time between the start of the emergency call and the pronunciation of the words "chest compressions," by the dispatcher
     * Median time elapsed between the start of the emergency call and the actual start of chest compressions by caller
     * Evaluation of the ventilation mode (hand on abdomen YES/NO, count the interval between two ventilatory movements YES/NO)
4. . Statistics

Sample size We need 100 patients in each period group to observe an absolute 20% difference in the rate of CA detection, compared with the detection rate of the control group (period 1) estimated at 60%, with an alpha risk = 0.05 and an 80% power in bilateral situations.

For each period:

- Description of patient characteristics and outcome

Comparison of these periods:

* Comparison of detection rate between the reference period (P1) and each of the other periods
* The number of subjects included in each period allows the realization of a χ² test with an alpha risk retained at 5%
* Adjust the detection rate on the significantly different variables between the groups (age, sex, no flow, time of rescuer arrival)
* The period 1 and 2 will be grouped and compared with period 3.

In all periods:

* Search variables associated with successful detection
* Multivariate logistic regression analysis type
* Survival analysis.
* Description of the evolution of the detection rate over time

ELIGIBILITY:
Inclusion Criteria:

Patient over 15 years old (adult morphology) suffering Out-of-hospital Cardiac Arrest before or during the call to the Dispatch Center

* Patient who benefited from the installation of a automated external defibrillator (AED) before or at the time of arrival of the rescuers on the scene

Exclusion Criteria:

Patient conscious at the time of the call

* OHCA between the end of the phone call and the arrival of rescuers on site
* OHCA after the rescuers' arrival on site
* Dispatch Center alerted on "second line" from another institution (Police, SAMU), without the possibility of joining the first caller.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: residents of Paris urban and suburban area
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Ratio of CA Detected by the emergency dispatcher | one year

SECONDARY OUTCOMES:
o Median time between the start of the emergency call and the pronunciation of the words "chest compressions," by the dispatcher | one year

OTHER OUTCOMES:
Median time elapsed between the start of the emergency call and the actual start of chest compressions by caller | one year
Evaluation of the ventilation mode (hand on abdomen YES/NO, count the interval between two ventilatory movements YES/NO) | one year
  , all calls related to Out -of-hospital Cardiac Arrest were registered , and in the days after, listened to and evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre TOURTIER, MDPhD Prof, Study Chair — Paris Fire Brigade - Emergency Medical Dept
Locations (1):
- Paris Fire Brigade Emergency Dept, Paris, France, France